CLINICAL TRIAL: NCT05627479
Title: Muscle Trauma, ATP Depletion, and Glucose-Insulin-Potassium Therapy (The MAGIK Trial): A Randomized, Controlled Feasibility Study of GIK Therapy to Decrease Skeletal Muscle Injury in Trauma Patients With Femoral Shaft (OTA 32A-C) and Tibial Shaft (OTA 42A-C) Fractures
Brief Title: MAGIK for Femoral/Tibial Shaft Fractures
Acronym: MAGIK
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to lack of funding.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01118
Record Dates: First submitted 2022-11-17; First posted 2022-11-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Femoral Shaft Fracture; Tibial Shaft Fracture
MeSH Terms: interventions — glucose-insulin-potassium cardioplegic solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GIK Therapy (Experimental): In patients randomized to the GIK Therapy Arm, a stepwise GIK infusion process will be performed. Baseline lab values that are markers of skeletal muscle injury (CPK), acute kidney injury (creatinine), and general tissue perfusion (lactate) will be obtained within the first 30 min of arrival to the ED. Subsequently, serial CPK, creatinine, myoglobin and lactate values will be obtained at regularly scheduled intervals until a minimum of 72 hours after definitive fixation or until rhabdomyolysis is resolved and/or kidney function has normalized
  Interventions: Drug: GIK solution
- Placebo Control (Placebo Comparator): Patients randomized to the control cohort will receive a normal saline infusion instead of GIK. Standard institutional ICU protocol will be used to monitor potassium and glucose levels per current standard-of-care practices and abnormal lab values will be treated accordingly per standard institutional protocols.
  Interventions: Drug: Isotonic Normal Saline Solution

INTERVENTIONS:
Drug: GIK solution — Therapy cocktail of Glucose, Insulin and Potassium. The medications will be prepared as per standard protocol. Administered intravenously.
  Arms: GIK Therapy
Drug: Isotonic Normal Saline Solution — Placebo injection - administered intravenously.
  Arms: Placebo Control

SUMMARY:
The purpose of this phase 2 randomized control trial will be to evaluate the effect of glucose-insulin-potassium (GIK) therapy in the setting of lower extremity trauma to reduce short- and long-term muscle damage, acute rhabdomyolysis, and acute kidney injury. The study will consist of 40 patients with femur or tibial shaft fractures randomized to the GIK arm (using a well-described systemic GIK protocol; n = 20) or the control arm (using isotonic saline; n = 20). The use of systemic GIK is expected to decrease the overall amount of lower extremity muscle cell death and result in improved muscle function in the postoperative period. Additionally, the investigators hypothesize that GIK will lead to less severe rhabdomyolysis and a concomitant decrease in the incidence of AKI that results from the byproducts of muscle cell death.

ELIGIBILITY:
Inclusion Criteria:

1. Femoral shaft fracture or tibial shaft fracture
2. Survival > 72 hours after definitive femur fracture fixation

Exclusion Criteria:

1. Pregnant women as the safety of GIK therapy in pregnant women has not been studied.
2. Age below 18 years
3. Survival < 72 hours after definitive femur fixation.
4. Pathologic fracture
5. Low energy bisphosphonate related atypical fracture
6. Patients with a contraindication to any of the medications on the study list
7. Patients with prior extremity weakness resulting from stroke or other neurological condition
8. Patients with absolute contraindications to undergoing MRI (implanted defibrillator or pacemaker, implanted deep brain stimulator, bullets or gunshot pellets near great vessels or vital organs, cerebral aneurysm clips, cochlear implants, magnetic dental implants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Peak Creatine Kinase (CK) Concentration During Hospital Stay | Up to Day 7 Post-Operation
  Measured via standard of care lab assessment.

SECONDARY OUTCOMES:
Number of Participants who Experience Acute Kidney Injury (AKI) | Up to Week 52 Post-Operation
Number of Participants with Stage 1 AKI | Up to Week 52 Post-Operation
Number of Participants with Stage 2 AKI | Up to Week 52 Post-Operation
Number of Participants with Stage 3 AKI | Up to Week 52 Post-Operation
Patient Reported Outcome Measurement Information System (PROMIS) Physical Function | Up to Week 52 Post-Operation
  Measure of self-reported capability rather than actual performance of physical activities. The raw score is the sum of responses and is calculated into a T-score with a mean of 50 and a standard deviation of 10; higher scores indicate greater physical function.
Quadriceps Muscle Strength in the Uninjured Leg | Up to Week 52
  Measured via handheld dynamometer.
Quadriceps Muscle Strength in the Injured Leg | Up to Week 52
  Measured via handheld dynamometer.
Hamstrings Muscle Strength in the Uninjured Leg | Up to Week 52
  Measured via handheld dynamometer.
Hamstrings Muscle Strength in the Injured Leg | Up to Week 52
  Measured via handheld dynamometer.
Uninjured Femur Muscle Volume at Week 4 Post-Op | Week 4 Post-Operation
  Muscle volume calculated via MRI.
Injured Femur Muscle Volume at Week 4 Post-Op | Week 4 Post-Operation
  Muscle volume calculated via MRI.
Uninjured Femur Muscle Volume at Week 24 Post-Op | Week 24 Post-Operation
  Muscle volume calculated via MRI.
Injured Femur Muscle Volume at Week 24 Post-Op | Week 24 Post-Operation
  Muscle volume calculated via MRI.
Uninjured Femur Muscle Volume at Week 52 Post-Op | Week 52 Post-Operation
  Muscle volume calculated via MRI.
Injured Femur Muscle Volume at Week 52 Post-Op | Week 52 Post-Operation
  Muscle volume calculated via MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit Konda, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [matthew.kingery@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be given access to the data upon reasonable request. Requests should be directed to matthew.kingery@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.